CLINICAL TRIAL: NCT06130163
Title: Benefits and Advantages of Intraoperative ERCP Versus Therapeutic Splitting in Cholecysto-, Choledocholithiasis in a High Expertise Center
Brief Title: Intraoperative ERCP Versus Therapeutic Splitting in Cholecysto-, Choledocholithiasis
Status: Completed | Type: Observational
Sponsor: Kepler University Hospital (Other)
Responsible Party: Principal Investigator, Dr. Sandra Raab, Dr. med. univ., Kepler University Hospital
Other Study IDs: ERCP
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2023-11

CONDITIONS: Cholelithiasis, Common Bile Duct
MeSH Terms: conditions — Choledocholithiasis | interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intraoperative ERCP: Patients with cholecystocholedocholithiasis getting intraoperative ERCP
  Interventions: Procedure: endoscopic retrograde cholangiopancreatography
- Splitting: Patients with cholecystocholedocholithiasis getting therapeutic splitting
  Interventions: Procedure: endoscopic retrograde cholangiopancreatography

INTERVENTIONS:
Procedure: endoscopic retrograde cholangiopancreatography — endoscopical clearance of the common bile duct
  Other Names: ERCP

SUMMARY:
At the Kepler University Hospital Linz all variants of ERCP (preoperative, intraoperative, postoperative ERCP) are performed in cases of simultaneous cholecysto- and choledocholithiasis. Hardly any other hospital in Austria prefers intraoperative ERCP or offers it at all. A standardized procedure with implemented logistics has been established. This study compares intraoperative and postoperative ERCP.

DETAILED DESCRIPTION:
At the Kepler University Hospital Linz all variants of ERCP (preoperative, intraoperative, postoperative ERCP) in cases of simultaneous cholecysto- and choledocholithiasis are performed. Usually an intraoperative ERCP followed by a preoperative ERCP is preferred. At the Kepler University hospital a high level of expertise in endoscopy and an interdisciplinary endoscopy team (surgical and internal medicine department) makes this high level of effort possible. Hardly any other hospital in Austria prefers intraoperative ERCP or offers it at all. A standardized procedure with implemented logistics has been established.

The aim of this study is to demonstrate and compare the advantages of both procedures at KUK from 1.1.2020 to 30.6.2023 (intraoperative and postoperative ERCP) in terms of morbidity, endoscopic success and the better way for patients and surgeons in clinics.

ELIGIBILITY:
Inclusion Criteria:

* simultaneous cholecysto-, choledocholithiasis
* emergency or elective
* confirmed choledocholithiasis
* intraoperative ERCP
* preoperative ERCP followed by cholecystectomy
* postoperative ERCP

Exclusion Criteria:

- < 18 years

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing surgery and ERCP in context to cholecysto-, choledocholithiasis in out hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Post-ERCP Pancreatitis | 48 hours after intervention
  radiological/blood sample/pain

SECONDARY OUTCOMES:
LOS | 9 months after first admission
  length of stay
Surgical method | at surgery
  LSK, robotic, open
Re-choledocholithiasis | up to one year after first admission
  choledocholithiasis after ERCP
Re-Intervenition | 30 days after surgery and/or ERCP
  any endoscopic/surgical/radiological intervention after surgery or ERCP
Successful ERCP | at ERCP
  yes or no
Costs | until 30 days after second surgery and/or ERCP
  costs for one patient

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Shamiyeh, Dr., Study Chair — Kepler University Hospital Linz; Sandra Raab, Dr., Principal Investigator — Kepler University Hospital Linz
Locations (1):
- Kepler University Hosital Linz, Linz, Austria, Austria